CLINICAL TRIAL: NCT00495664
Title: Titanium Nitride Oxide Coated Stents Versus Paclitaxel Eluting Stents for Acute Myocardial Infarction
Brief Title: Titanium Nitride Oxide Coated Stents and Paclitaxel Eluting Stents for Acute Myocardial Infarction
Acronym: TITAX AMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital District of Satakunta (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SA-002
Record Dates: First submitted 2007-07-02; First posted 2007-07-03 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2012-09

CONDITIONS: Acute Myocardial Infarction
Keywords: titanium; paclitaxel; stent; myocardial infarction; angioplasty; PCI
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TITANOX (Experimental): Titanium-nitride-oxide coated stent
  Interventions: Device: Titan stent and Taxus-Liberte stent
- PES (Active Comparator): Paclitaxel-eluting stent
  Interventions: Device: Titan stent and Taxus-Liberte stent

INTERVENTIONS:
Device: Titan stent and Taxus-Liberte stent

SUMMARY:
Coronary-stent implantation is commonly performed for treatment of acute myocardial infarction (MI). Drug eluting stents (DES) among selected patients have been shown to reduce target lesion revascularization (TLR) after percutaneous coronary intervention (PCI). However, there is no studies comparing titanium-nitride-oxide (TITANOX) coated stent with paclitaxel-eluting stent (PES) in acute MI.

DETAILED DESCRIPTION:
Study Design and Patient Population

The TITAX AMI (Titanium-Nitride-Oxide Coated stents versus Paclitaxel-Eluting Stents In Acute Myocardial Infarction) trial is a prospective, randomized and a multicenter trial conducted from December 2005 to November 2006 in six Finnish hospitals. The study was conducted according to the declaration of Helsinki and written informed consent was obtained from all patients. This protocol was approved by the Ethics Committees of the coordinating centre Satakunta Central Hospital and the participating hospitals.

Patients > 18 years of age presenting with acute MI (NSTEMI or STEMI) were eligible for this trial. Exclusion criteria included unprotected left main disease, ostial or restenotic lesions, contraindication to aspirin, clopidogrel or heparins, life expectancy of less than 12 months and if a stent longer than 28 mm was needed. According to the trial protocol, randomization was performed after visualization of the culprit lesion or a totally occluded infarct-related vessel during coronary angiography. Using sealed envelopes, patients were randomly assigned to the groups in a 1:1 ratio in each participating center.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age presenting with acute MI (NSTEMI or STEMI) were eligible for this trial.
* Wtitten informed consent

Exclusion Criteria:

* Restenosis
* Unprotected left main disease
* Ostial lesion
* Contraindication to asa, heparins, thienopyridines
* life expectancy < 12 months
* stent length needed > 28 mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2005-12; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
The primary end point was the first occurrence of major adverse cardiac event at 12 months defined as the composite of target lesion revascularization (TLR), recurrent MI, or death from cardiac causes. | One Year

SECONDARY OUTCOMES:
The secondary end points of the trial included all-cause mortality, composite of cardiac death or reinfarction and stent thrombosis. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Pasi Karjalainen, MD, Principal Investigator — Department of Cardiology, Satakunta Central Hospital
Locations (1):
- Satakunta Central Hospital, Pori, Finland

REFERENCES:
- [Derived] Karjalainen PP, Ylitalo A, Niemela M, Kervinen K, Makikallio T, Pietila M, Sia J, Tuomainen P, Nyman K, Airaksinen KE. Two-year follow-up after percutaneous coronary intervention with titanium-nitride-oxide-coated stents versus paclitaxel-eluting stents in acute myocardial infarction. Ann Med. 2009;41(8):599-607. doi: 10.1080/07853890903111018. PMID 19701826
- [Derived] Karjalainen PP, Ylitalo A, Niemela M, Kervinen K, Makikallio T, Pietili M, Sia J, Tuomainen P, Nyman K, Airaksinen KE. Titanium-nitride-oxide coated stents versus paclitaxel-eluting stents in acute myocardial infarction: a 12-months follow-up report from the TITAX AMI trial. EuroIntervention. 2008 Aug;4(2):234-41. doi: 10.4244/eijv4i2a42. PMID 19110789